CLINICAL TRIAL: NCT06367816
Title: Effectiveness, Safety and Efficacy of Closed-Loop Ventilation in Acute Brain Injury-Patients
Brief Title: Brain Recovery With Automated VEntilation
Acronym: BRAVE
Status: Recruiting | Type: Observational
Sponsor: University of Genova (Other)
Responsible Party: Principal Investigator, Lorenzo Ball, Clinical Professor, University of Genova
Other Study IDs: 13509
Record Dates: First submitted 2024-04-11; First posted 2024-04-16 (Actual); Last update posted 2024-05-02 (Actual); Status verified 2024-04

CONDITIONS: Brain Injuries, Acute; Respiration, Artificial; Automation
MeSH Terms: conditions — Brain Injuries; Respiratory Aspiration

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Procedure: INTELLiVENT — Closed-loop mode of ventilation
Procedure: Conventional ventilation — Mode of ventilation

SUMMARY:
Thus far, the closed-loop ventilation mode INTELLiVENT-ASV has been extensively tested in various groups of critically ill patients, and has been shown to be effective and safe in various groups of ventilated patients, including those at risk of acute respiratory distress syndrome (ARDS), patients with ARDS, and patients with chronic obstructive pulmonary disease (COPD). Some of these studies included acute brain injury (ABI) patients, but the effectiveness, efficacy and safety of INTELLiVENT-ASV has never been thoroughly tested in these patients. The current study will investigate the effectiveness in providing both brain- and lung protective ventilation, the safety and the efficacy of a closed-loop ventilation mode (INTELLiVENT-ASV) in acute brain injury patients, using breath-by-breath data.

DETAILED DESCRIPTION:
Rationale: Closed-loop ventilation has been proven effective in lung-protective ventilation but its effectiveness, safety and efficacy in providing both lung- and brain-protective ventilation in patients with acute brain injury has not been investigated.

Objective: To evaluate the effectiveness, efficacy and safety of INTELLiVENT-ASV with respect to brain- and lung-protective ventilation in ABI patients

Hypothesis: We hypothesize that INTELLiVENT-ASV is effective with regard to brain- and lung-protective ventilation (that is achieving brain- and lung- protective targets), efficacious (that is improving outcomes), and that INTELLiVENT-ASV is safe in invasively ventilated ABI patients.

Study design: Single-center, crossover trial.

Methods: In this prospective observational study, breath-by-breath ventilation data will be available from before and after the switch to closed-loop ventilation with INTELLiVENT-ASV, wherein the decision to switch is determined by the attending healthcare worker, i.e., not protocolized and only for clinical/organizational reasons. High granular data are collected both before and after this switch, limited to three hours for conventional and three hours for closed-loop ventilation. Neuromonitoring is part of current clinical practice and data will be collected only when available.

Study population: Invasively ventilated patients diagnosed with acute brain injury Methods: When the ventilator is switched upon the caregivers decision, data will be collected from three hours before the switch and three hours after the switch.

Study endpoints: The primary composite endpoint is the proportion of breaths and proportion of time within predefined zones of ventilation (based on VT and airway pressures, saturation of peripheral O2 (SpO2) and end-tidal CO2 (EtCO2).

ELIGIBILITY:
Inclusion Criteria:

* aged ≥ 18 years;
* intubated and receiving invasive ventilation for ABI;
* admitted to the Intensive Care Unit

Exclusion Criteria:

- receiving ventilation with a ventilator that does not allow INTELLiVENT-ASV

Ages: 18 Years to 105 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Invasively ventilated acute brain injury (ABI) patients admitted to the ICU of the Policlinico San Martino Hospital, Genova, Italy
Sampling Method: Non-Probability Sample
Enrollment: 20 (Estimated)
Dates: Start 2024-04-11 (Actual); Primary Completion 2024-12-31 (Estimated); Study Completion 2024-12-31 (Estimated)

PRIMARY OUTCOMES:
Proportion of breaths in predefined zones of ventilation | 7 hours from baseline
Proportion of time in predefined zones of ventilation | 7 hours from baseline

SECONDARY OUTCOMES:
Intracerebral changes assessed by multimodal neuromonitoring available | 7 hours from baseline
Changes on Electrical Impedence Tomography when available | 7 hours from baseline
Effectiveness in primary ABI patients vs non primary ABI patients | 7 hours from baseline
Episodes and time of high maximum airway pressure | 7 hours from baseline
Episodes and time of high respiratory rate | 7 hours from baseline
Incidence of severe hypoxemia | 7 hours from baseline
Incidence of severe hypercapnia | 7 hours from baseline
Discontinuation of ventilatory mode (yes or no) | 7 hours from baseline
Percentage of breaths in the predefined 'critical' ventilation zone | 7 hours from baseline
Incidence of pneumothorax | 8 hours from baseline
Efficacy on glascow coma scale | 7 hours from baseline
Duration of ventilation in survivors | 90 days
Ventilator free days | 90 days
Intensive care unit length of stay | 90 days
Hospital length of stay | 90 days
28-day mortality | 90 days
90-day mortality | 90 days
Number of alarms | 7 hours from baseline
Number of manual adjustments | 7 hours from baseline

CONTACTS AND LOCATIONS:
Locations (1):
- UO Clinica Anestesiologica e Terapia Intensiva, IRCCS Ospedale Policlinico San Martino, Genova, GE, Italy

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Goossen RL, Gavinelli S, Dragoni S, van Meenen DMP, Paulus F, Schultz MJS, Ball L, Patroniti NA, Robba C. Brain protective ventilation in acute brain injury patients with use of fully automated ventilation (BRAVE): A cross-over clinical trial. Eur J Anaesthesiol. 2025 Aug 25. doi: 10.1097/EJA.0000000000002253. Online ahead of print. PMID 40855946